CLINICAL TRIAL: NCT01332487
Title: Evaluating the Impact of Early Versus Delayed 5 Alpha Reductase Inhibitor Treatment on the Risk of Emergent Surgery in Men With Benign Prostatic Hyperplasia
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114461
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Results first posted 2012-02-29 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-05

CONDITIONS: Prostatic Hyperplasia
Keywords: 5-alpha-reductase inhibitor; prostate surgery; alpha-blocker; enlarged prostate; acute urinary retention; Benign prostatic hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Early initiation of 5ARI therapy: Patients starting 5ARI therapy within 30 days of initiating AB therapy
  Interventions: Drug: 5ARI + AB
- Delayed initiation of 5ARI therapy: Patients starting 5ARI therapy more than 30 days but less than 6 months from the initiation of AB therapy
  Interventions: Drug: 5ARI + AB

INTERVENTIONS:
Drug: 5ARI + AB — 5ARI: Dutasteride or Finasteride and any AB: Doxazosin, Prazosin, Tamsulosin, Terazosin or Alfuzosin

SUMMARY:
This retrospective study aims to assess the impact of early vs delayed 5-alpha-reductase inhibitor (5ARI) therapy in patients with BPH on alpha-blocker (AB) therapy and the risk of acute urinary retention (AUR), prostate-related surgery, and emergency surgery (defined as prostate surgery occurring within 30 days of AUR). The MarketScan database will be utilized for this study (2000-2008).

ELIGIBILITY:
Inclusion Criteria:

* Male
* aged 50 years or older
* diagnostic claim for BPH
* prescription claim for an AB and a 5ARI in the observation period (5ARI must occur within a 6-month window after the AB).
* continuously eligible for 6 months prior to and 12 months after index prescription date

Exclusion Criteria:

* prostate or bladder cancer during the study period
* any prostate-related surgical procedure within 5 months of the index prescription date
* prescription claim for finasteride 1 mg for male pattern baldness during the study period
* 5ARI therapy prior to initiation of AB therapy

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients aged 50 years or older with a diagnostic claim for BPH; prescription claim for an AB and a 5ARI in the observation period
Sampling Method: Probability Sample
Enrollment: 4068 (Actual)
Dates: Start 2010-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were neither recruited nor enrolled in this retrospective observational study. Data from medical records or insurance claims databases were anonymized.
Groups:
- Early Treatment: Participants who started 5-alpha-reductase inhibitor (5ARI) therapy within 30 days of initiating alpha-blocker (AB) treatment
- Delayed Treatment: Participants who started 5ARI therapy more than 30 days after initiating AB treatment but less than 6 months after initiating AB treatment
Period: Overall Study
Arm/Group | Early Treatment | Delayed Treatment
Started | 5554 | 3063
Completed | 5554 | 3063
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Early Treatment: Participants who started 5ARI therapy within 30 days of initiating AB treatment
- Total: Total of all reporting groups
Arm/Group | Early Treatment | Delayed Treatment | Total
Number analyzed (Participants) | 5554 | 3063 | 8617
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.7 (10.2) | 67.8 (10.1) | 68.4 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5554 | 3063 | 8617
Mean Charlson Comorbidity Index Scores [Mean (Standard Deviation); unit: scores on a scale] — The Charlson Comorbidity Index estimates 10-year mortality risk. Scores range from 0 - 37, with a lower score indicating a higher chance of survival.
  scores on a scale | 1.03 (1.63) | 0.86 (1.41) | 0.97 (1.56)
Mean Benign Prostatic Hyperplasia (BPH) Disease Stage Scores [Mean (Standard Deviation); unit: scores on a scale] — Disease staging for BPH was based on the International Classification of Diseases, 9th Revision (ICD-9), Clinical Modification codes. Scores: 0, BPH only; 1, BPH with urinary tract infection; 2, BPH with bladder outlet obstruction; 3, BPH with hydronephrosis; 4, BPH with renal failure; 5, BPH with sepsis; and 6, BPH with shock.
  scores on a scale | 0.90 (1.11) | 0.79 (0.98) | 0.86 (1.07)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Progression of Disease
Description: The number of participants in each study group with a treatment code for acute urinary retention, surgery, or emergency surgery (defined as surgery within 30 days following a diagnosis of acute urinary retention) was measured.
Time Frame: Up to 5 months
Population: Male participants age 50 years and older with a diagnosis of benign prostatic hyperplasia (BPH) or enlarged prostate (EP)
Measure: Number; unit: participants
Arm/Group | Early Treatment | Delayed Treatment
Number analyzed (Participants) | 5554 | 3063
participants
  Acute Urinary Retention | 589 | 393
  Surgery | 280 | 212
  Emergency Surgery | 86 | 52
Statistical Analysis 1: Comparison: Early Treatment vs Delayed Treatment; Test type: Superiority or Other; p = 0.002, Chi-squared — Acute Urinary Retention
Statistical Analysis 2: Comparison: Early Treatment vs Delayed Treatment; Test type: Superiority or Other; p = 0.000, Chi-squared — Surgery
Statistical Analysis 3: Comparison: Early Treatment vs Delayed Treatment; Test type: Superiority or Other; p = 0.597, Chi-squared — Emergency Surgery

2. Secondary Outcome: Number of Participants With the Indicated Time Between Acute Urinary Retention and Subsequent Surgery
Time Frame: 6 months
Population: Male participants age 50 years and older with a diagnosis of benign prostatic hyperplasia (BPH) or enlarged prostate (EP). Only those participants who were treated with surgery within 182 days of the first prescription of 5ARI were analyzed.
Measure: Number; unit: participants
Arm/Group | Early Treatment | Delayed Treatment
Number analyzed (Participants) | 106 | 68
participants
  On the same day | 37 | 27
  Within 1 week | 54 | 35
  Within 1 month | 85 | 51
  Within 2 months | 102 | 60
  Within 3 months | 105 | 64
  Within 4 months | 105 | 66
  Within 5 months | 105 | 68
  Within 6 months (182 days) | 106 | 68

ADVERSE EVENTS:
Description: This was a survey of participants, and adverse event/serious adverse event information was not captured in the study.
Arm/Group | Early Treatment | Delayed Treatment
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.